CLINICAL TRIAL: NCT07372066
Title: Effectiveness of Cognitive Stimulation Therapy Group for Residential Home Residents With Dementia and Mild Cognitive Impairment-- A Randomized Controlled Trial
Brief Title: Cognitive Stimulation Therapy Group for Residential Home Residents With Dementia and Mild Cognitive Impairment
Acronym: CSTSAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: The Hong Kong Society for the Aged (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-STA-00001945
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cognitive Functions
Keywords: Cognitive Stimulation Therapy; Calligraphy group; Randomized Controlled trial; Mild cognitive impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: This study adopts a multicentre randomized control trial two arms research design.
  The Cognitive Stimulation Therapy (CST) group provides weekly mental stimulation activities on a specific topic as mentioned above. It consists of a total of 14 sessions with two sessions per week, each lasting approximately 45 minutes and led by an occupational therapist. CST group consists of 14 sessions, with each session focusing on a theme, including: reality orientation, childhood, physical games, food, sound, faces, number games, word association, word games, current events, categorizing objects, using money, being creative, and team games. CST group will be delivered by trained occupational therapists.
  The Calligraphy group provides weekly calligraphy activities. It consists of a total of 14 sessions with two sessions per week, each lasting approximately 45 minutes and led by a rehabilitation assistant under the supervision of an occupational therapist.
Who Masked: Outcomes Assessor
Masking Description: A research staff, who does not involve in the group allocation and delivery of group interventions, conduct the intervention outcomes assessment of the participants before and after the intervention and 3-months follow-up. Standardized assessment tools are used to assess the intervention outcomes, including cognitive functions, depression, quality of life, and engagement and social functioning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive stimulation therapy (Active Comparator): In this study, the Cognitive Stimulation Therapy (CST) group follows the standard CST protocol of 14 sessions, with two sessions per week over a 7-week intervention period, as developed by Spector et al. (2003).
  Interventions: Behavioral: Cognitive Stimulation Therapy group
- Control group (Other): The control group participants will attend a calligraphy group consisting of 14 sessions, with two sessions per week. Each session will be led by a rehabilitation assistant under the supervision of an occupational therapist.
  Interventions: Behavioral: Calligraphy group

INTERVENTIONS:
Behavioral: Cognitive Stimulation Therapy group — The CST group provides weekly mental stimulation activities on a specific topic as mentioned above. It consists of a total of 14 sessions with two sessions per week, each lasting approximately 45 minutes and led by an occupational therapist. CST group consists of 14 sessions, with each session focusing on a theme, including: reality orientation, childhood, physical games, food, sound, faces, number games, word association, word games, current events, categorizing objects, using money, being creative, and team games. The stimulating activities are designed to match the abilities and interests of participants. CST groups will be delivered by trained occupational therapists.
  Arms: Cognitive stimulation therapy
Behavioral: Calligraphy group — The Calligraphy group offers weekly calligraphy activities, comprising 14 sessions in total, with two sessions per week. Each session lasts approximately 45 minutes and is led by a rehabilitation assistant under the supervision of an occupational therapist.
  Arms: Control group

SUMMARY:
The research aims to investigate the effectiveness a cognitive stimulation therapy group for older adults with dementia and mild cognitive impairment living in residential homes.

This study adopts a multicenter randomized control trial two arms research design. The randomized controlled trial will compare a typical 14-session cognitive stimulation therapy group with a calligraphy group to determine whether the 14-session cognitive stimulation therapy group can produce better intervention outcomes for older adults with dementia and mild cognitive impairment, including cognitive functions, depressive symptoms, activities engagement, social functioning and, quality of life.

DETAILED DESCRIPTION:
Objective: The research aims to investigate the effectiveness CST group for residential home residents with dementia and MCI. Additionally, the underlying mechanism of change of CST group will also be investigated.

Hypotheses.

1. The CST group is effective in improving cognitive abilities, depressive symptoms, engagement, social interaction and quality of life compared to the control group after the intervention.
2. The positive intervention results of the CST group are maintained at the 3-month follow-up
3. Improvement in cognitive ability is predicted by improved engagement in group activities.

Research Design. This study adopts a multicentre randomized control trial research design, involving 110 older people with dementia and MCI recruited from residential homes of SAGE. Using cluster randomization, participants will be openly recruited into activity groups in residential homes for older adults. The activity groups will then be randomly assigned to the intervention or control group in a 1:1 ratio. The intervention group will receive a 14-session CST group, while the control group will receive a calligraphy group. A research staff, who does not involve in the group allocation and group intervention, conduct the intervention outcomes assessment of the participants before and after the intervention and 3-months follow-up. Standardized assessment tools are used to assess the intervention outcomes, including cognitive functions, depression, quality of life, and engagement and social functioning. The ethical considerations of this study will be reviewed and approved by the Research Committee of the City University of Hong Kong. Data collection will begin in January 2026 and be completed in August 2026.

Subject Inclusion Criteria:

1. age 60 years or older;
2. diagnosis of MCI or dementia according to the Diagnostic and Statistical Manual of Mental Disorder (Fifth edition, Text Revision); Participants who do not receive a diagnosis of MCI or dementia will undergo a screening assessment by a researcher using the Chinese Montreal Cognitive Assessment (MoCA)-5 minutes.

Subject Exclusion Criteria Those who are unable to participate independently in group activities, who exhibit disruptive behavior and/or are severely impaired by physical disabilities (e.g. severe hearing and visual impairment) and physical illnesses (e.g. frequent hospital stays) are excluded.

Sample size estimation. The sample size of this study is estimated by using power analysis G*Power 3.1. Recent studies on CST suggest a medium to large effect size on improving cognitive function. This study aims to detect a medium effect size (i.e., Cohen's d = 0.40) with a statistical power of 0.80 for all intervention outcomes and with a dropout rate of 20%, 110 people with dementia will be recruited in this study.

Intervention and Control Group Activities. The participants are randomly assigned to an intervention group or a control group. The intervention group receives the Cognitive Simulation Therapy (CST) group, while the control group receives the calligraphy group.

The CST group provides weekly mental stimulation activities on a specific topic as mentioned above. It consists of a total of 14 sessions with two sessions per week, each lasting approximately 45 minutes and led by an occupational therapist. CST group consists of 14 sessions, with each session focusing on a theme, including: reality orientation, childhood, physical games, food, sound, faces, number games, word association, word games, current events, categorizing objects, using money, being creative, and team games. The stimulating activities are designed to match the abilities and interests of participants.

The Calligraphy group provides weekly calligraphy activities. It consists of a total of 14 sessions with two sessions per week, each lasting approximately 45 minutes and led by a rehabilitation assistant under the supervision of an occupational therapist.

Outcomes Assessment Tools The primary intervention outcome of this study is the improvement of cognitive ability as measured by the Chinese Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) and the Chinese Montreal Cognitive Assessment (MoCA), which have been used as outcome assessment in previous studies of Chinese older adults with MCI.

The secondary intervention outcomes of this study are the improvement in depressive symptoms, engagement, social interaction and quality of life which are assessed by the following standardized scales.

* The Chinese Cornell Scale for Depression in Dementia (CSDD) is a 19-item scale for assessing the mood changes in older adults with dementia and MCI rated by the caregivers.
* The Chinese Quality of Life-Alzheimer's disease (QoL-AD) is a 13item scale for assessing the QoL in older adults with dementia and MCI. In this study, QoL-AD is completed by both older adults with dementia and MCI as well as their caregivers independently to give self-rated and caregiver-rated QoL.
* The Engagement of a person with dementia scale (EPWDS) is a 10-item scale to assess five areas of engagement in in older adults with dementia and MCI, including affect, visual, verbal, behavioural and social, rated by the caregivers.
* The Chinese Social Functioning in Dementia scale (SF-DEM) is a 20-item scale for assessing social interactions with family, friends, and the community in older adults with dementia and MCI. In the present study, the SF-DEM is completed by both older adults with dementia and MCI as well as their caregivers independently to give self-rated and caregiver-rated social functioning.
* The Clinical Sustainability Assessment Tool (CSAT) is a 35-item scale for assessing the sustainability of clinical practices for the intervention group. This scale is rated by management and professional staff of SAGE residential homes.

Data Analyses. The analysis is carried out according to the intent-to-treat principle, whereby the multiple imputation method is used for missing data. The data analyses are performed with SPSS 29.0. Within-group intervention effects will be analyzed for all intervention groups using repeated measures one-way analysis of variance (ANOVA). Between group intervention effects are analyzed using 2 (group) x 2 (time) repeated measures of ANOVA. Within and between group effect sizes are computed using Cohen's d, with values of 0.2, 0.5, and 0.8 considered as small, medium, and large respectively.

Fidelity of intervention. Standardized program manuals for CST group and calligraphy group will be designed by the research team to suit the needs and interests of participants with dementia and MCI. The occupational therapists conducting the CST group have completed training on conducting CST group. In addition, they receive the standardized program manuals, training and regular supervision, as well as a surprise check from the research team when conducting the CST group to ensure that the interventions implemented by the occupational therapists meet the guidelines and skills of the standardized program manuals. The rehabilitation assistant conducting the calligraphy group will receive the standardized program manuals, training and regular supervision by an occupational therapist to ensure that the interventions conducted by rehabilitation assistant meet the guidelines and skills of the standardized program manuals.

Ethical Considerations. The ethical aspects of this study were reviewed and approved by the Research Committee of the City University of Hong Kong [Reference No.: HU-STA-00001945]. Written informed consent will be obtained from all participants and their guardians on the day of the screening before participants start receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age 60 years or older;
2. diagnosis of MCI or dementia according to the Diagnostic and Statistical Manual of Mental Disorder (Fifth edition, Text Revision).

Remark: Participants who do not receive a diagnosis of MCI or dementia will undergo a screening assessment by a researcher using the Chinese Montreal Cognitive Assessment (MoCA)-5 minutes.

Exclusion Criteria:

Those who are unable to participate independently in group activities, who exhibit disruptive behavior and/or are severely impaired by physical disabilities (e.g. severe hearing and visual impairment) and physical illnesses (e.g. frequent hospital stays) are excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog | ADSA_cog will be used before intervention, after 7 weeks intervention, and 3-month follow-up.
  The ADAS-Cog has good validity and internal consistency (Cronbach's α = 0.9; Chu et al., 2000), and covers eleven cognitive tasks, including word recall, naming objects and fingers, commands, constructional praxis, ideational praxis, orientation, word recognition, language, comprehension of spoken language, and word finding difficulty. Total scores range from 0 to 70, with higher scores signify more severe cognitive impairment.
MoCA | MoCA will be used before intervention, after 7 weeks intervention, and 3-month follow-up.
  The MoCA has satisfactory validity, internal consistency (Cronbach's α = 0.8; Yeung et al., 2014), and is widely used for screening and assessment of mild cognitive impiarment (Chen et al, 2021). It assesses global and specific cognitive abilities, including memory recall, attention, concentration, executive functions, language, visuospatial skills, abstract reasoning, calculation and orientation (Yeung et al., 2014). The scores are summed over the items, with a total score ranginge from 1 to 30. Higher scores indicate better cognitive abilities.

SECONDARY OUTCOMES:
Chinese Cornell Scale for Depression in Dementia (CSDD) | CSDD will be used before intervention, after 7 weeks intervention, and 3-month follow-up.
  The Chinese Cornell Scale for Depression in Dementia (CSDD) is a 19-item scale for assessing the mood changes in older adults with dementia and MCI rated by the caregivers with satisfactory validity and internal consistency (Cronbach's α = 0.82; Lin et al., 2008). Each item (e.g., lack of reaction to pleasure) is rated using a 3-point scale: absent (0), mild or intermittent (1), and severe (2). The scores are summed across the items, with a total score ranging from 0 to 38. Higher scores indicate greater severity of depressive symptoms.
Chinese Quality of Life-Alzheimer's disease (QoL-AD) | QoL-AD will be used before intervention, after 7 weeks intervention, and 3-month follow-up.
  The Chinese Quality of Life-Alzheimer's disease (QoL-AD) is a 13 item scale for assessing the QoL in older adults with dementia and MCI, with satisfactory validity and internal consistency (Cronbach's α = 0.78 to 0.92; Chan et al., 2009). In the present study, the QoL-AD scale is completed by both older adults with dementia and MCI as well as their caregivers independently to give self-rated and caregiver-rated QoL. Each item (e.g. "How do you feel about your physical health?") is rated on a 4-point scale (poor = 1, fair = 2, good = 3, excellent = 4). The scores are summed across the items, yielding a total score ranging from 13 to 52. Higher scores indicate better quality of life.
Engagement of a person with dementia scale (EPWDS) | EPWDS will be used before intervention, after 7 weeks intervention, and 3-month follow-up
  The Engagement of a person with dementia scale (EPWDS) is a 10-item scale to assess five areas of engagement in in older adults with dementia and MCI, including affect, visual, verbal, behavioural and social, rated by the caregivers with satisfactory validity and good internal consistency (Cronbach's α = 0.94; Jones et al., 2018). Each item (e.g. displays positive affect such as pleasure, contentment or excitement) is rated on a 5-point Likert scale, with scores ranging from "1" (strongly agree) to "5" (strongly disagree). The scores are summed across the items, with a total score ranging from 10 to 50. Higher scores indicate a higher level of positive engagement.
The Chinese Social Functioning in Dementia scale (SF-DEM) | It will be used before the intervention, after 7-weeks intervention and 3-months follow-up.
  The Chinese Social Functioning in Dementia scale (SF-DEM) is a 17-item scale for assessing social interactions with family, friends, and the community in older adults with dementia and MCI, with acceptable validity and internal consistency (Cronbach's α = 0.60 to 0.64; Chan et al., 2009). In the present study, the SF-DEM is completed by both older adults with dementia and MCI as well as their caregivers independently to give self-rated and caregiver-rated social functioning. Each item (e.g. Asked other people about their feelings or concerns) is rated using a 4-point scale, ranging from "0" (never) to "3" (always). The scores are summed over the items, with a total score raning from 0 to 51. Higher scores indicate better social functioning.
Clinical Sustainability Assessment Tool (CSAT) | It will be used after 7-weeks intervention
  The Clinical Sustainability Assessment Tool (CSAT) is a 35-item scale for assessing the sustainability of clinical practices for the intervention group, with acceptable validity and internal consistency (Cronbach's α = 0.91; Malone et al., 2021). This scale is rated by management and professional staff of SAGE residential homes. CAST assesses seven domains, including engaged staff and leadership, engaged stakeholders, organisational readiness, workflow integration, implementation and training, monitoring and evaluation, and outcomes and effectiveness. Each domain consists of five items. Each item is rated using a 7-point Likert scale, ranging from "1" (none) to "7" (highest). The scores for each domain are summed across the items, with a total score ranging from 1 to 35. Higher scores indicate greater capacity and sustainability.

CONTACTS AND LOCATIONS:
Locations (1):
- SAGE Old Age Homes, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woods B, Rai HK, Elliott E, Aguirre E, Orrell M, Spector A. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2023 Jan 31;1(1):CD005562. doi: 10.1002/14651858.CD005562.pub3. PMID 39804128
- [Background] Wong A, Yiu S, Nasreddine Z, Leung KT, Lau A, Soo YOY, Wong LK, Mok V. Validity and reliability of two alternate versions of the Montreal Cognitive Assessment (Hong Kong version) for screening of Mild Neurocognitive Disorder. PLoS One. 2018 May 23;13(5):e0196344. doi: 10.1371/journal.pone.0196344. eCollection 2018. PMID 29791452
- [Background] Thorgrimsen L, Selwood A, Spector A, Royan L, de Madariaga Lopez M, Woods RT, Orrell M. Whose quality of life is it anyway? The validity and reliability of the Quality of Life-Alzheimer's Disease (QoL-AD) scale. Alzheimer Dis Assoc Disord. 2003 Oct-Dec;17(4):201-8. doi: 10.1097/00002093-200310000-00002. PMID 14657783
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Malone S, Prewitt K, Hackett R, Lin JC, McKay V, Walsh-Bailey C, Luke DA. The Clinical Sustainability Assessment Tool: measuring organizational capacity to promote sustainability in healthcare. Implement Sci Commun. 2021 Jul 17;2(1):77. doi: 10.1186/s43058-021-00181-2. PMID 34274004
- [Background] Gomez-Soria I, Iguacel I, Aguilar-Latorre A, Peralta-Marrupe P, Latorre E, Zaldivar JNC, Calatayud E. Cognitive stimulation and cognitive results in older adults: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2023 Jan;104:104807. doi: 10.1016/j.archger.2022.104807. Epub 2022 Sep 6. PMID 36116285
- [Background] Desai R, Leung WG, Fearn C, John A, Stott J, Spector A. Effectiveness of Cognitive Stimulation Therapy (CST) for mild to moderate dementia: A systematic literature review and meta-analysis of randomised control trials using the original CST protocol. Ageing Res Rev. 2024 Jun;97:102312. doi: 10.1016/j.arr.2024.102312. Epub 2024 Apr 16. PMID 38636561
- [Background] Chen X. Effectiveness of cognitive stimulation therapy (CST) on cognition, quality of life and neuropsychiatric symptoms for patients living with dementia: A meta-analysis. Geriatr Nurs. 2022 Sep-Oct;47:201-210. doi: 10.1016/j.gerinurse.2022.07.012. Epub 2022 Aug 6. PMID 35940038
- [Background] Cao Y, Wang N, Zhang Q, Shen N, Bai J, Luo X, Liu Y. Effects of cognitive stimulation therapy on patients with dementia: An umbrella review of systematic reviews and meta-analyses. Exp Gerontol. 2023 Jun 15;177:112197. doi: 10.1016/j.exger.2023.112197. Epub 2023 May 6. PMID 37146891
- [Background] Davis LC, Diianni AT, Drumheller SR, Elansary NN, D'Ambrozio GN, Herrawi F, Piper BJ, Cosgrove L. Undisclosed financial conflicts of interest in DSM-5-TR: cross sectional analysis. BMJ. 2024 Jan 10;384:e076902. doi: 10.1136/bmj-2023-076902. PMID 38199616